CLINICAL TRIAL: NCT06362538
Title: Cardiovascular Prevention Program at Maria Cecilia Hospital
Brief Title: The Cardiovascular Prevention Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Cecilia Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: MCH-ProCardioPrev
Record Dates: First submitted 2024-03-20; First posted 2024-04-12 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-03

CONDITIONS: Cardiovascular Prevention
MeSH Terms: interventions — Carotid Intima-Media Thickness; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- subject with a negative or positive history of cardiovascular disease (Other): no drugs or devices are included.
  Interventions: Other: International Physical Activity Questionnaire; Other: Six minute walking test; Other: SF-36, Euro-Qol 5D-5L, Perceived stress scale-10, Pittsburgh Sleep Quality Index, Depression Anxiety Stress scale- 21.; Other: MEDAS; Other: Intima-media thickness (IMT); Biological: Blood sampling; Biological: Stool Sample Culture Test

INTERVENTIONS:
Other: International Physical Activity Questionnaire — Assessments of physical activity level and functional capabilities (aerobic capacity, muscular strength and power, flexibility
Other: Six minute walking test — The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Other: SF-36, Euro-Qol 5D-5L, Perceived stress scale-10, Pittsburgh Sleep Quality Index, Depression Anxiety Stress scale- 21. — Evaluation of the quality of life, the psychological sphere (anxiety, stress, depression) and the quality of sleep
Other: MEDAS — Evaluation of adherence to the Mediterranean diet
Other: Intima-media thickness (IMT) — Bmode ultrasonography
Biological: Blood sampling — Measurement of parameters for defining cardiovascular risk and biomarkers.
Biological: Stool Sample Culture Test — Evaluation of Gut Microbiota

SUMMARY:
Cardiovascular diseases represent one of the main public health problems being the leading cause of morbidity, disability and mortality. In recent decades, the global prevalence and cardiovascular disease mortality has increased, with 23.6 million annual deaths expected by 2030. In Europe, mortality per year is equal to 2.2 million women and 1.9 million men, representing 47% and 37% of all deaths respectively. In Italy, the situation in terms of deaths due to cardiovascular diseases it is in line with the world ranking and European, being responsible for 44% of all deaths. The only interventional or pharmacological approach is neither effective nor sustainable. The most deaths from cardiovascular diseases are due to atherothrombotic events, which are attributable to a series of risk factors, most of which are modifiable. Turns out itself as a targeted action on these factors with the aim of safeguarding the state of health cardiovascular, may represent the best applicable strategy. It is therefore necessary structure and activate prevention programs aimed at the general population and groups of subjects at higher risk.

ELIGIBILITY:
Inclusion Criteria:

* primary prevention: age ≥ 30 years with a negative history of cardiovascular events
* secondary prevention: age ≥ 30 years with a negative history of cardiovascular events

Exclusion Criteria:

* severe obesity
* high-grade renal failure
* severe and/or dialysis
* oncological disease in active phase
* pregnancy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
measure of body mass index | 12 months
  BMI Assessment
Adherence to the Mediterranean diet | 12 months
  Mediterranean Diet Adherence
blood test to check cholesterol levels | 12 months
  Assessment of hypercholesterolemia
blood pressure measurement | 12 months
  Evaluation of Diastolic Blood Pressure
blood glucose test | 12 months
  evaluation of blood glucose

CONTACTS AND LOCATIONS:
Overall Officials: Anna Maria Malagoni, Principal Investigator — Maria Cecilia Hospital
Locations (1):
- MCH, Cotignola, Ravenna, Italy

IPD SHARING:
Plan to Share IPD: No